CLINICAL TRIAL: NCT04657575
Title: Optimisation of Electro-Convusions-Therapie (ECT) Based on ASTI (Anaesthesia to Intervention Time Interval) Versus Narcotrend - a Randomised Prosepctive
Brief Title: Optimisation of ECT Based on ASTI vs Narcotrend
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ECT: ASTI vs Narcotrend
Record Dates: First submitted 2020-11-23; First posted 2020-12-08 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2022-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASTI (No Intervention): ECT guided with ASTi 2-4 min
- Narcotrend (Active Comparator): ECT guided with ECT
  Interventions: Procedure: Narcotrend

INTERVENTIONS:
Procedure: Narcotrend — ECT stimulation within an anaesthesia depth range of 41-64
  Arms: Narcotrend

SUMMARY:
The Electro-Convulsion-Therapy (ECT) is a well accepted treatment option in severe depression. The quality of ECT is evaluated basing on minimal seizure duration (>15sec), the sympathic response and the postictal EEG-suppression.

- Page 1 of 3 - For the treatment general anaesthesia is needed. On the other hand anaesthesia strongly influences the quality of the seizure. Standard treatment is to use Anaesthesia to intervention time (ASTI) of 1 to 2 minutes for ideal timing of the electric stimulation.

The aim of the study is to assess if timing of electric stimulation aiming for ar an anaesthesia depth of Narcotrend values 41-64 may provide better convulsion quality than standard approach of using ASTI 1-2 minutes.

DETAILED DESCRIPTION:
The Electro-Convulsion-Therapy (ECT) is a well accepted treatment option in severe depression. The quality of ECT is evaluated basing on minimal seizure duration (>15sec), the sympathic response and the postictal EEG-suppression.

- Page 1 of 3 - For the treatment general anaesthesia is needed. On the other hand anaesthesia strongly influences the quality of the seizure. Standard treatment is to use Anaesthesia to intervention time (ASTI) of 1 to 2 minutes for ideal timing of the electric stimulation.

The aim of the study is to assess if timing of electric stimulation aiming for ar an anaesthesia depth of Narcotrend values 41-64 may provide better convulsion quality than standard approach of using ASTI 1-2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Age: 18 -90 years
* Signed informed consent
* Severe depressive disorder

Exclusion Criteria:

* ASA >3
* Age < 18 or > 90
* denial of the patient
* Impossibility to fix Narcotrend electrodes
* Patients unable to consent
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Convulsion Quality | One hour
  Adequate seizure quality was defined as > 20 seconds motor response on the right forearm, >25 seconds EEG seizure activity, postictal suppression index > 80%, maximum sustained coherence > 90% and 5.midictal amplitude > 180µV

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Hospital Innsbruck, Innsbruck, Tyrol, Austria